CLINICAL TRIAL: NCT01025232
Title: A Phase I/II Open Label, Multicenter Study of the Safety, Tolerability and Efficacy of Multiple Intravitreal Injections of (Super-dose Anti-VEgf SAVE Trial) 2.0mg Ranibizumab in Subjects With Chronic Fluid on OCT Post Multiple Injections With Ranibizumab
Brief Title: A Study of Intravitreal Injections of 2.0mg Ranibizumab in Subjects With Chronic Fluid On OCT Post Multiple Injections With Ranibizumab (Super-dose Anti-VEgf SAVE Trial)
Acronym: SAVE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The last remaining subject withdrew consent because the collaborator Genentech stopped supplying study drug.
Sponsor: David M. Brown, M.D. (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, David M. Brown, M.D., Director Of Research, Greater Houston Retina Research
Organization: Greater Houston Retina Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FVF4571s
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Results first posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-11

CONDITIONS: Age Related Macular Degeneration; Choroidal Neovascular Membrane; Subfoveal Neovascular Age-Related Macular Degeneration; Macular Degeneration; Wet Age-Related Macular Degeneration
Keywords: Antibodies, Monoclonal; Immunologic Factors; Eye Diseases; Retinal Degeneration; Macular Degeneration; Pharmacologic Actions; Retinal Diseases
MeSH Terms: conditions — Macular Degeneration; Eye Diseases; Retinal Degeneration; Retinal Diseases | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4 Week Re-treatment (Active Comparator): Subjects can receive re-treatment every 4 weeks if there is persistent or recurrent intraretinal, subretinal, or sub-RPE fluid on any OCT modality, or any evidence of hemorrhage on clinical evaluation. Subjects will go no longer than 12 weeks without treatment.
  Interventions: Drug: Ranibizumab
- 6 Week Re-treatment (Active Comparator): Subjects can receive re-treatment every 6 weeks if there is persistent or recurrent intraretinal, subretinal, or sub-RPE fluid on any OCT modality, or any evidence of hemorrhage on clinical evaluation. Every 6 weeks regimen will test potential longer duration of action of 2.0 mg ranibizumab. Subjects will go no longer than 12 weeks without treatment.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal Injection of 2.0mg formulation
  Other Names: Lucentis

SUMMARY:
The purpose of this study is to determine whether 2.0mg Ranibizumab is effective in the treatment of recurrent fluid.

DETAILED DESCRIPTION:
This is an open-label, Phase I/II study of intravitreally administered 2.0 mg ranibizumab in subjects with persistent fluid or recurrent fluid on OCT after having received at least nine ranibizumab injections in the past twelve months. Consented, enrolled subjects will receive have monthly ETDRS BCVA, ophthalmic examination and OCTs evaluation using Stratus, Cirrus and Spectralis machines. Fluorescein angiography and autofluorescence will be done at BSL, and Months 6 and 12. DNA samples for genetic analysis will be collected at baseline.

Subjects will receive open-label intravitreal injections of 2.0 mg ranibizumab administered every 28 days for 3 months: Following the three loading doses, all patients will receive a minimum "capped" PRN treatment (all patients will receive 2.0 mg intravitreal ranibizumab quarterly). Dosing should not occur earlier than 22 days after the previous treatment. Study visits should be scheduled to occur every 30 (±7) days relative to the date of the first injection (Day 0).

Subjects will be randomized into two re-treatment cohorts for additional re-treatment, if needed:

* Cohort A - Subjects can receive re-treatment every 4 weeks if there is persistent or recurrent intraretinal, subretinal ,or sub-RPE fluid on any OCT modality, or any evidence of hemorrhage on clinical evaluation.
* Cohort B - Subjects can receive re-treatment every 6 weeks if there is persistent or recurrent intraretinal, subretinal ,or sub-RPE fluid on any OCT modality, or any evidence of hemorrhage on clinical evaluation. Every 6 weeks regimen will test potential longer duration of action of 2.0 mg ranibizumab.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to provide signed informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization
* Age ≥ 50 years
* For sexually active women of childbearing potential, agreement to the use of an appropriate form of contraception (or abstinence) for the duration of the study
* Although no birth control method is 100% effective, the following are considered effective means of contraception: surgical sterilization, use of oral contraceptives, barrier contraception using either a condom or diaphragm with spermicidal gel, an intrauterine device, or contraceptive hormone implant or patch. A patient's primary care physician, obstetrician, or gynecologist should be consulted regarding an appropriate form of birth control.
* Ability and willingness to return for all scheduled visits and assessments

Study eyes must meet the following criteria for entry into the SAVE trial:

* The last treatment with Ranibizumab is ≥ 28 days
* To have received at least 9 injections of Ranibizumab in the past 12 months
* Any CNVM lesion (Occult, Minimally Classic or Classic) (i.e., leakage on fluorescein angiography or subretinal, intraretinal, or sub-RPE fluid on Spectral Domain OCT) secondary to age-related macular degeneration.
* Best corrected visual acuity in the study eye, using e-ETDRS testing, between 20/25 and 20/320 (Snellen equivalent), inclusive.
* Only one eye will be enrolled in the Study. If both eyes are eligible study investigator will select the eye for entry.
* The total area of subretinal hemorrhage and fibrosis must comprise less than 50% of the total lesion.
* Clear ocular media and adequate pupillary dilation to permit good quality fundus imaging

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or lactation Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial

Ocular Exclusion Criteria Prior Ocular Treatment

* History of vitrectomy surgery, submacular surgery, or other surgical intervention for AMD in the study eye
* Prior treatment with Visudyne®, external-beam radiation therapy, or transpupillary thermotherapy (TTT) in the study eye at a fluence equal to 100%, any fluence lower than 100% is permitted.
* Prior treatment with full or half fluence verteporfin PDT.
* Previous intravitreal drug delivery (e.g., intravitreal corticosteroid injection, anti-angiogenic drugs besides ranibizumab, or device implantation) in the study eye within the last 12 months.

CNV Lesion Exclusion Characteristics

* Subretinal hemorrhage in the study eye that involves the center of the fovea, if the size of the hemorrhage is either > 50% of the total area of the lesion or > 1 disc area (2.54 mm2) in size
* Subfoveal fibrosis or atrophy in the study eye
* CNV in either eye due to other causes, such as ocular histoplasmosis, trauma, or pathologic myopia Concurrent Ocular Conditions
* Retinal pigment epithelial tear involving the fovea in the study eye
* Any concurrent intraocular condition in the study eye (e.g., cataract or diabetic retinopathy) that, in the opinion of the investigator, could either:

Require medical or surgical intervention during the 24-month study period to prevent or treat visual loss that might result from that condition; or If allowed to progress untreated, could likely contribute to loss of at least 2 Snellen equivalent lines of BCVA over the 24-month study period.

* Active intraocular inflammation (grade trace or above) in the study eye
* Current vitreous hemorrhage in the study eye
* History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Aphakia or absence of the posterior capsule in the study eye
* Intraocular surgery (including cataract surgery) in the study eye within 2 months preceding Day 0
* Uncontrolled glaucoma in the study eye (defined as IOP ≥ 30 mmHg despite treatment with anti-glaucoma medication)
* History of glaucoma-filtering surgery in the study eye
* History of corneal transplant in the study eye

Concurrent Systemic Conditions (Exclusion)

* Uncontrolled blood pressure (defined as systolic > 180 mmHg and/or diastolic > 110 mmHg while patient is sitting) If a patient's initial reading exceeds these values, a second reading may be taken 30 or more minutes later. If the patient's blood pressure needs to be controlled by antihypertensive medication, the patient can become eligible if medication is taken continuously for at least 30 days prior to Day 0.
* Atrial fibrillation not managed by patient's primary care physician or cardiologist within 3 months of screening visit
* Women of childbearing potential not using adequate contraception (as defined in the inclusion criteria).

A woman is considered not to be of childbearing potential if she is postmenopausal, defined by amenorrhea for at least 1 year in a woman > 45 years old; or has undergone hysterectomy and/or bilateral oophorectomy.

* History of stroke within the last 3 months of screening visit
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug or that might affect interpretation of the results of the study or renders the patient at high risk for treatment complications
* Current treatment for active systemic infection
* Active malignancy
* History of allergy to fluorescein, not amenable to treatment
* Inability to obtain fundus photographs or fluorescein angiograms of sufficient quality to be analyzed and graded by the central reading center
* Inability to comply with study or follow-up procedures
* Previous participation in any studies of investigational drugs within 1 month preceding Day 0 (excluding vitamins and minerals)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2009-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Brown, MD, Principal Investigator — Greater Houston Retina Research
Locations (2):
- United States (2):
  - Greater Houston Retina Research, Houston, Texas
  - Greater Houston Retina Research, The Woodlands, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 4 Week Re-treatment | 6 Week Re-treatment
Started | 46 | 42
Completed | 43 | 36
Not Completed | 3 | 6
Not completed — Study drug no longer available | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4 Week Re-treatment | 6 Week Re-treatment | Total
Number analyzed (Participants) | 46 | 42 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 44 | 39 | 83
Age, Continuous [Mean (Full Range); unit: years] | 76 [60 to 93] | 77 [53 to 87] | 76.1 [53 to 93]
Gender [Count of Participants; unit: Participants]
  Female | 25 | 21 | 46
  Male | 21 | 21 | 42
Region of Enrollment [Number; unit: participants]
  United States | 46 | 42 | 88

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in ETDRS BCVA at Month 12 (Fixed Interval Dosing Primary Endpoint After 3 Monthly Doses. Variable Interval Dosing Primary Endpoint at 1 Year.)
Description: Early Treatment Diabetic Retinopathy Study Best Corrected Visual Acuity (ETDRS BCVA) was used to quantify visual acuity. BCVA is measured using an eye chart and is reported as the number of letters read correctly using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved.
Time Frame: 1 Year
Measure: Mean (Standard Error); unit: ETDRS BCVA Letters
Arm/Group | 4 Week Re-treatment | 6 Week Re-treatment
Number analyzed (Participants) | 43 | 36
ETDRS BCVA Letters | 4.1 (1.4) | 4.1 (1.0)

2. Secondary Outcome: Evaluate the Incidence and Severity of Ocular and Non-ocular Adverse Events (AEs) Through Month 12
Time Frame: 1 year
Measure: Number; unit: Incidents
Arm/Group | 4 Week Re-treatment | 6 Week Re-treatment
Number analyzed (Participants) | 46 | 42
Incidents
  Ocular Events | 18 | 8
  Serious Non-Ocular Events | 7 | 10

3. Secondary Outcome: Determine Number of Patients Who Experience a Loss of 15 or More Letters From Baseline to Month 12 and Month 12 in ETDRS BCVA
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | 4 Week Re-treatment | 6 Week Re-treatment
Number analyzed (Participants) | 46 | 42
participants | 1 | 0

4. Secondary Outcome: Determine Number of Patients Who Experience a Gain of 15 or More Letters From Baseline to Month 12 in ETDRS BCVA.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | 4 Week Re-treatment | 6 Week Re-treatment
Number analyzed (Participants) | 46 | 42
participants | 5 | 3

5. Secondary Outcome: Evaluate Mean Change in Central Retinal Thickness Over Time Through Month12 as Assessed by All Three OCTs (Stratus, Cirrus, and Spectralis)
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | 4 Week Re-treatment | 6 Week Re-treatment
Number analyzed (Participants) | 46 | 42
micrometer | -59.2 (107.8) | -31.8 (87.2)

6. Secondary Outcome: Assess Number of Ranibizumab Injections in Each of the Two Doses Required Through Month 12
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: number of injection
Arm/Group | 4 Week Re-treatment | 6 Week Re-treatment
Number analyzed (Participants) | 46 | 42
number of injection | 11.6 (1.1) | 8.6 (0.8)

7. Secondary Outcome: Evaluate the Relationship Between Specific Genetic Polymorphisms Associated With AMD, Disease Characteristics and Processes, and Response to Intravitreal Ranibizumab
Time Frame: 1 year
Population: Given lack of clinical benefit of 2.0 mg ranibizumab, as demonstrated in the HARBOR trial [Busbee BG, et al. (2013) Ophthalmology 120(5), 1046-1056], further secondary analyses were suspended.
Arm/Group | 4 Week Re-treatment | 6 Week Re-treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | 4 Week Re-treatment | 6 Week Re-treatment
Serious Adverse Events (participants affected / at risk) | 7/46 | 10/42
Other Adverse Events (participants affected / at risk) | 18/46 | 8/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 4 Week Re-treatment (N=46) | 6 Week Re-treatment (N=42)
Death (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 1
Idiopathic internal bleeding (Blood and lymphatic system disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pancreatic cancer (Hepatobiliary disorders) | 1 | 2
Lung cancer (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 | 2
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 4 Week Re-treatment (N=46) | 6 Week Re-treatment (N=42)
RPE rip (Eye disorders) | 0 | 1
Subretinal hemorrhage (Eye disorders) | 3 | 2
Vitreous hemorrhage (Eye disorders) | 1 | 1
Vein occlusion (Eye disorders) | 1 | 0
Increase in NS (Eye disorders) | 3 | 0
Increase in PSC (Eye disorders) | 4 | 0
Cataract surgery (Eye disorders) | 3 | 0
PVD (Eye disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes